CLINICAL TRIAL: NCT06219564
Title: Diagnostic Accuracy of MRI to Predict Peripartum Hysterectomy and Neonatal Mortality in Total Placenta Previa: A Retrospective Cohort Study.
Brief Title: Total Placenta Previa Associated With the Placenta Accreta Spectrum.
Acronym: PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sadık Kükrer, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SBU-OBGYN-SK-01
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Maternal; Procedure
Keywords: magnetic resonance imaging; obstetric labor complications; placenta percreta; placenta previa; pregnancy complications
MeSH Terms: conditions — Obstetric Labor Complications; Placenta Accreta; Placenta Previa; Pregnancy Complications | interventions — Cesarean Section; Infant Mortality

STUDY DESIGN:
Intervention Model Description: 277 singleton pregnancies that met the inclusion criteria and were diagnosed with total placenta previa (t-PP) in the third trimester were divided into two groups according to whether a placental-MRI (p-MRI) was performed. Nevertheless, we explored whether pregnant women diagnosed with total placenta previa (t-PP), with or without a placental-MRI (p-MRI), needed to undergo peripartum-total abdominal hysterectomy (p-TAH) during cesarean section (C/S) due to the placenta accreta spectrum (PAS).
Who Masked: Outcomes Assessor
Masking Description: Two radiologists with at least ten years of experience, independently of each other, evaluated p-MRI scans of pregnant women diagnosed with t-PP without prior knowledge of the original reports.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total placenta previa (t-PP) patients who underwent placental MRI (p-MRI). (Active Comparator): The study compares clinical factors and p-MRI findings between two surgical procedures: Caesarean Section (C/S) and Peripartum Total Abdominal Hysterectomy (p-TAH). The study analyzes both univariate and multivariate associations with surgical procedures.
  This arm presents the results of a study assessing risk factors affecting peripartum hysterectomy in placenta previa patients, focusing on the impact of MRI screening. Peripartum hysterectomy (p-TAH) refers to the surgical removal of the uterus around the time of childbirth.
  The arm does not explicitly mention specific interventions to be administered. However, it provides information on clinical and p-MRI factors that might influence the surgical procedure (C/S or p-TAH) choice in placenta previa patients. The interventions, if any, would likely be based on assessing these risk factors and involve decisions on the type of surgery, additional procedures, or use of certain medical interventions based on the patient's condition.
  Interventions: Procedure: Peripartum total abdominal hysterectomy (p-TAH); Procedure: Cesarean Section (C/S); Other: Neonatal mortality
- Total placenta previa (t-PP) patients who did not undergo placental MRI (p-MRI). (Active Comparator): The study compares clinical factors without p-MRI between two surgical procedures: Cesarean Section (C/S) and Peripartum Total Abdominal Hysterectomy (p-TAH). The study analyzes both univariate and multivariate associations with surgical procedures.
  This arm presents the results of a study assessing risk factors affecting peripartum hysterectomy (p-TAH) in placenta previa patients, focusing on the impact of clinical factors.
  The arm does not explicitly mention specific interventions to be administered. However, it provides information on clinical factors that might influence the surgical procedure (C/S or p-TAH) choice in placenta previa patients. The interventions, if any, would likely be based on assessing these risk factors and involve decisions on the type of surgery, additional procedures, or use of certain medical interventions based on the patient's condition.
  Interventions: Procedure: Peripartum total abdominal hysterectomy (p-TAH); Procedure: Cesarean Section (C/S); Other: Neonatal mortality

INTERVENTIONS:
Procedure: Peripartum total abdominal hysterectomy (p-TAH) — Peripartum total abdominal hysterectomy (cesarean hysterectomy) refers to a surgical procedure in which a woman undergoes both a cesarean section (C-section) and a hysterectomy simultaneously.
  Placenta Accreta, Increta, or Percreta: These are conditions where the placenta attaches too deeply to the uterine wall. In cases of severe attachment, it may be difficult to remove the placenta without causing excessive bleeding, and a hysterectomy may be required.
  Cesarean hysterectomy is a major surgical procedure involving significant medical expertise and coordination among healthcare professionals, including obstetricians and surgeons. The decision to perform a cesarean hysterectomy is usually made in emergency situations to address life-threatening complications.
  Other Names: Cesarean hysterectomy
Procedure: Cesarean Section (C/S) — A cesarean section (C/S) involves making an incision in the abdominal wall and uterus to deliver a baby when a vaginal delivery is not feasible or safe.
  Total placenta previa refers to a condition where the placenta completely covers the opening of the cervix in the uterus. This condition can pose significant risks during pregnancy and childbirth, and it often necessitates a planned cesarean section (C/S) for delivery.
  Other Names: C-section
Other: Neonatal mortality — Neonatal mortality refers to the death of a newborn within the first 28 days of life. This period is divided into early neonatal mortality, which covers the first seven days of life, and late neonatal mortality, which extends from the eighth to the 28th day. Neonatal mortality is a critical measure of the health and well-being of infants and is often used to assess a population's overall health and healthcare systems.
  To reduce neonatal mortality, efforts are made to improve maternal healthcare, access to prenatal care, skilled attendance during childbirth, and the availability of neonatal healthcare services. Tracking and addressing factors contributing to neonatal mortality are crucial for improving the chances of survival of newborns and overall health outcomes.

SUMMARY:
To assess the reliability of placental magnetic resonance imaging measurements in predicting peripartum hysterectomy and neonatal outcomes in patients with total placenta previa.

DETAILED DESCRIPTION:
Study design and patients This study analyzed the outcomes of a cohort of 372 pregnant women diagnosed with PP over five years, from November 2017 to June 2023. The patient population for the study included women between the ages of 17 and 42 who were in their third trimester of pregnancy (27th to 37th weeks of gestation) and had received a t-PP diagnosis via color Doppler ultrasonography (cd-USG) and/or p-MRI. The resulting cohort compared a final sample population of 277 singleton pregnant women with t-PP, which comprised 150 pregnant women who underwent antenatal p-MRI examinations in the third trimester and 127 pregnant women who did not undergo a p-MRI.

Standards of reference The study covered all singleton pregnancies in which t-PP extended to both the anterior and posterior uterine walls, resulting in complete coverage of the internal cervical os by the placenta. Transvaginal and transabdominal USG were planned between 32 and 34 weeks for all patients who were followed up in our clinic due to t-PP and were scheduled to be delivered. The gestational ages of the participants were determined using the last menstrual date and crown-rump length (CRL) measurements from a first-trimester ultrasound. Two perinatologists with at least ten years of experience examined each patient's cd-USG for signs of PAS. Ultrasonographic signs identified included placental lacunae, placenta previa involving the cervix, loss of the clear zone, and bladder wall interruption.

Two radiologists with at least ten years of experience, independently of each other, evaluated p-MRI scans of pregnant women diagnosed with t-PP without prior knowledge of the original reports.

Definitive diagnosis and pathological reporting Pathological reports and approvals were granted according to a rigorous protocol involving at least two pathologists, each with a minimum of seven years of professional expertise in their field.

p-MRI image interpretations The assessment focused on analyzing the different positions of the atypical placenta in the lower uterine segment, including the anterior, posterior, anterolateral, and posterolateral locations. Precise measurements were taken to calculate the placental volume in the S1 and S2 sectors, cervical canal length, and cervical canal dilatation. Based on sagittal p-MRI scans, the placental invasion was classified into two main areas. Implementing a plane perpendicular to the upper bladder's axis facilitated the boundary of these sectors. The term S1 refers to the upper uterine segment that forms the part of the uterus that contacts the bladder's posterior wall. Likewise, the lower uterine segment, identified as S2, was formed in the lower posterior wall of the bladder. Radiologists conducted a sector-wise (S1 and S2) examination of the invasion topography, which allowed them to identify specific invasion locations, including parametrial and cervical involvement and bladder interruption.

Multidisciplinary team The operations of patients who gave birth due to PAS were performed by the same multidisciplinary team, which included perinatologists, gynecological and obstetric surgeons, gynecological oncologists, urologists, neonatologists, cardiovascular surgeons, anesthesiology and reanimation specialists, interventional radiologists, and allied health personnel with ten years of experience.

Scheduled surgery and preoperative preparations All participants in our study underwent cesarean births during the third trimester of pregnancy. Except for urgent situations, all scheduled preterm cesarean deliveries and p-TAH procedures were conducted during the gestational period of 34+0 to 36+6 weeks. Among the patients admitted to our clinic due to t-PP, surgical intervention was performed before the planned delivery date in cases of uterine contraction, the onset of vaginal bleeding, or unexpected medical indications for the mother and fetus.

Statistical Method and Power Analysis G*Power V. 3.1.9.6 estimated sample size. All p-MRI values of patients with and without PAS were compared in the reference study, and the difference was substantial. Using 95% confidence (1-α), 95% test power (1-β), d=0.8 effect size, and the two-way hypothesis, the study contained 84 cases, with a minimum of 42 in each group. The study included 155 cesarean sections and 122 TAH cases; post hoc analysis revealed a power of 99.9%. 16 Data were analyzed using IBM SPSS V23. ROC analysis determined the surgical procedure variable cut-off values. Univariate and multivariate binary logistic regression analyses examined independent surgical risk factors. Backward-Wald method was used for multivariate binary logistic regression. The analysis findings present mean ± standard deviation, median (minimum-maximum), and frequency (percentage) for quantitative and categorical variables. Intraclass correlation coefficients and Kappa (k) tests were conducted to assess intra- and inter-observer agreement reliability. The significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 27th to 37th weeks of gestation
* Third trimester of pregnancy
* Pregnants had received a t-PP diagnosis via color Doppler ultrasonography (cd-USG) and/or placental MRI (p-MRI).
* All singleton pregnancies in which t-PP extended to both the anterior and posterior uterine walls, resulting in complete coverage of the internal cervical os by the placenta

Exclusion Criteria:

* Any cases of low-lying/marginal placenta previa
* Preoperative hemoglobin level < 9 g/dL
* Pregnant women with coagulation disorders
* Morbid obesity
* Multiple fetal pregnancies
* Individuals delivered before < 27 weeks of gestation

Ages: 17 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — singleton pregnant women
Enrollment: 277 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of risk factors affecting peripartum hysterectomy in placenta previa patients undergoing without MRI screening | Assessed during the peripartum period, within the first two days postpartum.
  Binary measure indicating whether peripartum hysterectomy occurred (yes/no).
Clinical risk factors affecting p-TAH in patients with t-PP undergoing p-MRI. | Assessed during the peripartum period, within the first 2 days postpartum.
  Binary measure indicating whether peripartum hysterectomy occurred (yes/no).
Identification of risk factors affecting neonatal mortality regardless of whether MRI scanning is used. | Assessed at the time of delivery.
  Binary measure indicating whether neonatal mortality occurred (yes/no).

SECONDARY OUTCOMES:
The ROC analysis of the placental volume (S1 and S2 sectors), CCL, and CCD obtained from the p-MRI scan for indications of peripartum hysterectomy | Assessed based on ROC analysis.
  Assessment of the ability of different variables (S1, S2, CCL, CCD) to indicate the need for peripartum hysterectomy.
Peripartum Hysterectomy Occurrence | Assessed during the peripartum period, within the first 2 days postpartum.
  1. Participants and Procedures:
     * Two surgery procedures are compared: Cesarean Section (C/S) and Total Abdominal Hysterectomy (TAH).
     * The participants are divided into those who underwent C/S (155 cases) and TAH (122 cases).
  2. Risk factors that could potentially impact surgery type:
     * Age of the mother
     * Prior D&C procedure
     * Previous C-section delivery
     * Vaginal delivery without complications
     * Past myomectomy surgery
     * Hysteroscopy procedure
     * Weeks of gestational age
     * Antepartum hemorrhage
     * Fetal birth weight
     * Blood product transfusions
     * MRI screenings (S1, S2, CCL, CCD)

CONTACTS AND LOCATIONS:
Overall Officials: Sadık Kükrer, Principal Investigator — SBU Adana Training and Research Hospital, Department of Obstetrics and Gynecology, Adana, Turkey; Sefa Arlıer, Study Chair — SBU Adana Training and Research Hospital, Department of Obstetrics and Gynecology, Adana, Turkey; Okan Dilek, Study Chair — SBU Adana Training and Research Hospital, Department of Radiology, Adana, Turkey; Çağrı Gülümser, Study Director — Yuksek Ihtisas University, Department of Obstetrics and Gynecology, Ankara, Turkey; Işıl Adıgüzel, Study Chair — SBU Adana Training and Research Hospital, Department of Obstetrics and Gynecology, Adana, Turkey
Locations (1):
- University of Health Sciences Adana City Training and Research Hospital, Department of Obstetrics and Gynecology, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huijgen QC, Gijsen AF, Hink E, Van Kesteren PJ. Cervical tourniquet in case of uncontrollable haemorrhage during caesarean section owing to a placenta accreta. BMJ Case Rep. 2013 Apr 22;2013:bcr2013009237. doi: 10.1136/bcr-2013-009237. PMID 23608864
- [Result] Jha P, Poder L, Bourgioti C, Bharwani N, Lewis S, Kamath A, Nougaret S, Soyer P, Weston M, Castillo RP, Kido A, Forstner R, Masselli G. Society of Abdominal Radiology (SAR) and European Society of Urogenital Radiology (ESUR) joint consensus statement for MR imaging of placenta accreta spectrum disorders. Eur Radiol. 2020 May;30(5):2604-2615. doi: 10.1007/s00330-019-06617-7. Epub 2020 Feb 10. PMID 32040730
- [Result] Morel O, Collins SL, Uzan-Augui J, Masselli G, Duan J, Chabot-Lecoanet AC, Braun T, Langhoff-Roos J, Soyer P, Chantraine F; International Society for Abnormally Invasive Placenta (IS-AIP). A proposal for standardized magnetic resonance imaging (MRI) descriptors of abnormally invasive placenta (AIP) - From the International Society for AIP. Diagn Interv Imaging. 2019 Jun;100(6):319-325. doi: 10.1016/j.diii.2019.02.004. Epub 2019 Mar 8. PMID 30853416
- [Result] Palacios Jaraquemada JM, Bruno CH. Magnetic resonance imaging in 300 cases of placenta accreta: surgical correlation of new findings. Acta Obstet Gynecol Scand. 2005 Aug;84(8):716-24. doi: 10.1111/j.0001-6349.2005.00832.x. PMID 16026395
- [Result] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Result] Jauniaux E, Hussein AM, Fox KA, Collins SL. New evidence-based diagnostic and management strategies for placenta accreta spectrum disorders. Best Pract Res Clin Obstet Gynaecol. 2019 Nov;61:75-88. doi: 10.1016/j.bpobgyn.2019.04.006. Epub 2019 Apr 30. PMID 31126811
- [Result] Hecht JL, Baergen R, Ernst LM, Katzman PJ, Jacques SM, Jauniaux E, Khong TY, Metlay LA, Poder L, Qureshi F, Rabban JT 3rd, Roberts DJ, Shainker S, Heller DS. Classification and reporting guidelines for the pathology diagnosis of placenta accreta spectrum (PAS) disorders: recommendations from an expert panel. Mod Pathol. 2020 Dec;33(12):2382-2396. doi: 10.1038/s41379-020-0569-1. Epub 2020 May 15. PMID 32415266
- [Result] Hobson SR, Kingdom JC, Murji A, Windrim RC, Carvalho JCA, Singh SS, Ziegler C, Birch C, Frecker E, Lim K, Cargill Y, Allen LM. No. 383-Screening, Diagnosis, and Management of Placenta Accreta Spectrum Disorders. J Obstet Gynaecol Can. 2019 Jul;41(7):1035-1049. doi: 10.1016/j.jogc.2018.12.004. PMID 31227057
- [Result] Romeo V, Verde F, Sarno L, Migliorini S, Petretta M, Mainenti PP, D'Armiento M, Guida M, Brunetti A, Maurea S. Prediction of placenta accreta spectrum in patients with placenta previa using clinical risk factors, ultrasound and magnetic resonance imaging findings. Radiol Med. 2021 Sep;126(9):1216-1225. doi: 10.1007/s11547-021-01348-6. Epub 2021 Jun 22. PMID 34156592
- [Result] Jauniaux E, Bhide A, Kennedy A, Woodward P, Hubinont C, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Prenatal diagnosis and screening. Int J Gynaecol Obstet. 2018 Mar;140(3):274-280. doi: 10.1002/ijgo.12408. No abstract available. PMID 29405319
- [Result] Chen X, Shan R, Song Q, Wei X, Liu W, Wang G. Placenta percreta evaluated by MRI: correlation with maternal morbidity. Arch Gynecol Obstet. 2020 Mar;301(3):851-857. doi: 10.1007/s00404-019-05420-5. Epub 2020 Jan 4. PMID 31903499
- [Result] Gulati A, Anand R, Aggarwal K, Agarwal S, Tomer S. Ultrasound as a Sole Modality for Prenatal Diagnosis of Placenta Accreta Spectrum: Potentialities and Pitfalls. Indian J Radiol Imaging. 2021 Oct 19;31(3):527-538. doi: 10.1055/s-0041-1735864. eCollection 2021 Jul. PMID 34790294
- [Result] Bhide A, Laoreti A, Kaelin Agten A, Papageorghiou A, Khalil A, Uprichard J, Thilaganathan B, Chandraharan E. Lower uterine segment placental thickness in women with abnormally invasive placenta. Acta Obstet Gynecol Scand. 2019 Jan;98(1):95-100. doi: 10.1111/aogs.13422. Epub 2018 Aug 2. PMID 29978457
- [Result] Elmaraghy AM, Taha Fayed S, Abd ElHamid Ali M, Ali Hassanien M, Mohamed Mamdouh A. Diagnostic Accuracy of Placental Thickness in Lower Uterine Segment Measured by Ultrasound in Prediction of Placenta Accreta Spectrum in Patients with Placenta Previa. A Diagnostic Test Accuracy Study. Int J Womens Health. 2023 Feb 16;15:311-320. doi: 10.2147/IJWH.S399520. eCollection 2023. PMID 36814526
- [Result] Takahashi H, Matsubara S. Placental thickness measurement is difficult in some cases. Acta Obstet Gynecol Scand. 2019 Feb;98(2):264-265. doi: 10.1111/aogs.13443. Epub 2018 Sep 12. No abstract available. PMID 30129148
- [Result] Altal OF, Qudsieh S, Ben-Sadon A, Hatamleh A, Bataineh A, Halalsheh O, Amarin Z. Cervical tourniquet during cesarean section to reduce bleeding in morbidly adherent placenta: a pilot study. Future Sci OA. 2022 Mar 8;8(4):FSO789. doi: 10.2144/fsoa-2021-0087. eCollection 2022 Apr. PMID 35369280
- [Result] Matsuzaki S, Nagase Y, Takiuchi T, Kakigano A, Mimura K, Lee M, Matsuzaki S, Ueda Y, Tomimatsu T, Endo M, Kimura T. Antenatal diagnosis of placenta accreta spectrum after in vitro fertilization-embryo transfer: a systematic review and meta-analysis. Sci Rep. 2021 Apr 28;11(1):9205. doi: 10.1038/s41598-021-88551-7. PMID 33911134
- [Result] Salmanian B, Fox KA, Arian SE, Erfani H, Clark SL, Aagaard KM, Detlefs SE, Aalipour S, Espinoza J, Nassr AA, Gibbons WE, Shamshirsaz AA, Belfort MA, Shamshirsaz AA. In vitro fertilization as an independent risk factor for placenta accreta spectrum. Am J Obstet Gynecol. 2020 Oct;223(4):568.e1-568.e5. doi: 10.1016/j.ajog.2020.04.026. Epub 2020 Apr 30. PMID 32360847
- [Result] Vermey BG, Buchanan A, Chambers GM, Kolibianakis EM, Bosdou J, Chapman MG, Venetis CA. Are singleton pregnancies after assisted reproduction technology (ART) associated with a higher risk of placental anomalies compared with non-ART singleton pregnancies? A systematic review and meta-analysis. BJOG. 2019 Jan;126(2):209-218. doi: 10.1111/1471-0528.15227. Epub 2018 May 8. PMID 29740927
- [Result] Imafuku H, Tanimura K, Shi Y, Uchida A, Deguchi M, Terai Y. Clinical factors associated with a placenta accreta spectrum. Placenta. 2021 Sep 1;112:180-184. doi: 10.1016/j.placenta.2021.08.001. Epub 2021 Aug 5. PMID 34375912